CLINICAL TRIAL: NCT06295445
Title: Impact of Integrated Cardiopulmonary Ultrasound on Clinical Outcome of Shocked Patients in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Cardiopulmonary Ultrasound
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Shock
MeSH Terms: conditions — Shock | interventions — Caves; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Control group (Experimental): About 54 patients that will undergo treatment without any use of point of care cardio-pulmonary ultrasound scans for guidance of the management.
  Interventions: Other: treatment without any use of point of care cardio-pulmonary ultrasound scans for guidance of the management
- Group B: Study group (Experimental): About 54 patients that will undergo cardio-pulmonary ultrasound guided management.
  Interventions: Procedure: care cardio-pulmonary ultrasound

INTERVENTIONS:
Procedure: care cardio-pulmonary ultrasound — Evaluation of the heart and lung conditions in shocked patients using focused cardio-pulmonary ultrasound for treatment guidance and their implication on the patient's outcome
  Other Names: Echo
  Arms: Group B: Study group
Other: treatment without any use of point of care cardio-pulmonary ultrasound scans for guidance of the management — treatment without any use of point of care cardio-pulmonary ultrasound scans for guidance of the management
  Arms: Group A: Control group

SUMMARY:
Shock is one of the most common conditions in the intensive care unit (ICU) affecting one-third of critically ill patients. It reduces oxygen and nutrition's perfusion to the solid organs and is closely associated with increased mortality. Most literature has described how hemodynamic monitoring could provide an effective way to identify underlying pathophysiological processes and guide appropriate therapy in shock patients.

DETAILED DESCRIPTION:
The diagnosis of shock is based on clinical, hemodynamic, and biochemical signs. It is manifested with systemic arterial hypotension with mean arterial pressure less than 70 mm Hg, with reflex tachycardia. Also, there are clinical signs of tissue hypoperfusion, including cutaneous hypoperfusion with cold clammy skin, renal hypoperfusion with resulting oliguria (urine output [UOP] <0.5 ml/kg/h) and neurologic hypoperfusion with altered mental state. Tissue hypoperfusion leads to anaerobic tissue metabolism with hyperlactatemia (>1.5 mmol/L).

Assessment of hemodynamic status and lines of management of the acute circulatory shock remains a challenging issue in emergency medicine and critical care. As the use of invasive hemodynamic monitoring declines, bedside-focused ultrasound (US) has become a valuable tool in the evaluation and management of patients in shock.

Four types of shock exist, including hypovolemic, cardiogenic, distributive, and obstructive shock. Clinical assessment and classification of shock is extremely difficult in critically ill patients as there is sometimes an overlap between these types. Incorporation of bedside ultrasound in patients with undifferentiated shock allows for rapid evaluation of reversible causes of shock and improves accurate diagnosis in undifferentiated hypotension.

Currently, the critical care ultrasound (CCUS) has been widely advocated as the preferred tool to assess hemodynamics, including accurately estimating pathophysiological changes of shock. This information, therefore, can be carried out into protocols to guide shock treatment. However, despite previous recommendations, current protocols are subjective and empirical, without listing specific variables as indicators, such as ejection fraction (EF), mitral annular plane systolic excursion (MAPSE), tricuspid annular plane systolic excursion (TAPSE),mitral or tricuspid annular peak systolic velocity (S'-MV or S'-TV), inferior vena cava (IVC), and lung ultrasound score (LUSS).

CCUS examination on ICU admission which performed by the experienced physician provide valuable information to assist the caregivers in understanding the comprehensive outlook of the characteristics of hemodynamics and lung pathology. Those key variables obtained by CCUS predict the possible prognosis of patients, hence deserve more attention in clinical decision making.

Lung ultrasound has been widely used in diagnosing pulmonary diseases including pneumonia, connective tissue diseases and interstitial lung diseases. For patients in the intensive care unit (ICU), more attention is paid to monitoring the development of lung pathologic changes, which guides the therapy. Lung insults caused by inflammation, trauma or water increase always lead to infiltration, which results in the loss of lung air. Depending on the severity of the aeration loss and water increase, each part of the lung generates different ultrasound signs upon exam.

The lung ultrasound score (LUSS) is the sum of the scores of each exam zone and has been justified as a respectable semiquantitative score to measure the lung aeration loss caused by different lung pathologic changes, such as pneumonia, atelectasis, pleural effusion, and lung edema.

Lung Ultrasound Protocol (LUSS): Reliable techniques have been used based on the international evidence-based recommendations for point-of-care lung ultrasound that recommended using a complete eight-zone lung ultrasound examination to evaluate the LUSS. The anterior and lateral chest wall are divided into eight areas. Areas 1 and 2 denote the upper anterior and lower anterior chest areas, respectively, and areas 3 and 4 denote the upper lateral and basal lateral chest areas, respectively.

ELIGIBILITY:
Inclusion Criteria:

* state of hypotension represented by systolic BP <90 mm Hg or mean arterial pressure (MAP) <60 mmHg).
* serum lactate level of ≥ 2 mmol/L
* positive with at least one of the conditions below: Lactate level >2mmol/L.
* Capillary Refill Time >4.5s; Urine output per hour <0.5ml/kg; Clammy skin, limbs cold. unconsciousness. initiation of intravenous vasopressors .

Exclusion Criteria:

* Patients with trauma history,
* Patients with suspected or diagnosed raised intra-abdominal or intrathoracic pressures as pregnancy, Portal hypertension, Mediastinal mass, Intracerebral hemorrhage, Increased intracranial pressure, Valvular heart disease,Atrial fibrillation.
* Patients or families refused to participate in the study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 72 hours of the initial fluid resuscitation
  Time of mortality occurrence since randomization, comparing intervention and control group.
Number of mortalities | 72 hours of the initial fluid resuscitation
  Amount of non-survivor subject, comparing intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hussein Fahmy, Professor, Study Chair — Anesthesia, Intensive Care and Pain Management Department,Al-Azhar University, Faculty of medicine for boys; Moaz Atef El-Shahat, Lecturer, Study Director — Chest Diseases Department,Al-Azhar Faculty of Medicine; Hani Abdelshafook, Lecturer, Principal Investigator — Cardiology Department, Al-Azhar Faculty of Medicine
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No